CLINICAL TRIAL: NCT00117221
Title: MRI Measurement of Brain Metabolism Across the Sleep-Wake Cycle
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050179; 05-N-0179
Record Dates: First submitted 2005-07-02; First posted 2005-07-04 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2014-02-11

CONDITIONS: Sleep
Keywords: Magnetic Resonance Imaging; Functional Imaging; Cerebral Blood Flow; BOLD Effect; Sleep

SUMMARY:
This study will investigate the spatio-temporal characteristics of brain activity during sleep. Functional magnetic resonance imaging (fMRI) studies have shown that in the absence of external stimuli, the brain continues to show spatial patterns of activity that resemble those during sensory and cognitive tasks. This phenomenon greatly affects the interpretation of neuroimaging studies based on positive emission tomography (PET) and fMRI, which rely on the contrast between brain activity during a task and activity during rest. In addition, resting state activity in itself may reveal information on the large-scale organization of neuronal networks and on functional abnormalities related to disease.

Participants should represent a broad cross section of the healthy adult population. Any neurologically and psychiatrically healthy male or nonpregnant female between 18 and 65 years old may be eligible.

Studies will be conducted in the In Vivo NMR Research Center. Concurrent electroencephalogram (EEG) and MRI studies will last between 1 and 2 hours. A typical study involves 15 minutes of anatomical MRI scanning followed by a 60-minute functional scan during which the subject relaxes with eyes closed and is encouraged to sleep while the fMRI/EEG are performed. Participants may be scanned 1 to 20 times. No more than 1 scan will be performed per day and no more than 20 scans will be performed within a year. During the last 5 to 10 minutes of the scan, the participant will open his or her eyes and actively participate in a visual stimulation or attention task. The participant's alertness will be measured by a behavioral (button-press) response. The visual stimuli (contrast reversing checkerboard displays, alternated with uniform grey fields) will be presented using the standard projection system available with the MRI scanner. The attention task will involve repeated visual presentation of groups of letters and digits; the participant will be asked about the correspondence between these groups.

Magnetoencephalogram (MEG) scans will be performed on some participants. The precise and undistorted signals available with MEG will be used to enhance the interpretation of alertness and sleep-related characteristics of the EEG signals, which can vary quite dramatically across subjects. In addition, the MEG signals will provide preliminary spatial localization of the sleep-dependent changes more precisely than is possible with EEG. MRI scanner noise will be simulated using tape recordings to allow comparison with the MRI/EEG data. MEG scans will last 45 minutes to 2 hours. At all times during any of the brain scans the participant will be able to communicate the MRI scientist or MEG/EEG technician and can ask to be removed from the device at any time.

The study will not have a direct benefit for participants. It may be help us learn more about brain function, which may lead to better treatments.

DETAILED DESCRIPTION:
Objective. The objective of the proposed study is to investigate the spatio-temporal characteristics of brain activity during sleep. A number of recent fMRI (Ogawa, Lee et al. 1990) studies have shown that in absence of external stimuli, the brain continues to show spatial patterns of activity that resemble the networks that activate during sensory and cognitive tasks. This phenomenon greatly affects the interpretation of neuroimaging studies based on PET and fMRI, since these rely on differential imaging in which activity during a task is contrasted against activity during rest. In addition, resting state activity in itself potentially contains unique information on the large scale organization of neuronal networks and reveals information about functional abnormalities related to disease processes.

Study Population. To avoid confounding factors related to disease processes, subjects for this study will be recruited from the normal adult population. In addition, subjects will be screened for sleep behavior, and subjects with abnormal sleep behavior will be excluded.

Design. The study is designed to facilitate MRI detection of cerebral metabolic differences between the sleep and awake states. Wakefulness and sleep, and the various stages will be classified in accordance with the EEG criteria, consistent with the guidelines of Rechtschaffen and Kales (Rechtschaffen, 1968). For this purpose, we will optimize the methodology for the concurrent acquisition of EEG and fMRI signals. Using concurrent EEG and state-of-the-art MRI, we plan to establish the precise spatial distribution of changes in brain activity that are associated with changes in the sleep/wake state and the various stages of sleep, specifically early sleep (stage 1 and 2). Secondly, we plan to investigate whether changes in regional brain metabolism as measured by MRI correlates with transitory EEG phenomena during sleep, including fluctuations in band-specific power, sleep spindles, and K-complexes.

Outcome Measure. As an outcome of this study, an atlas of activity clusters in normal subjects will be established, both during waking conditions, as well as during several sleep stages. Further outcomes will be spatial patterns of covariance with EEG band-specific power, spindles, and K-complexes. These data will serve as a baseline for comparison with activity patterns in patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any neurologically and psychiatrically normal, male or female, healthy volunteer between 18 and 65 years old is in principle eligible for the study. Subjects must be capable of understanding the procedures and requirements of this study. Subjects must be willing to sign an informed consent document.

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contraindication to MR scanning such as the following: pregnancy, aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; known absent acoustic reflex; ocular foreign body (e.g. metal shavings or insulin pump) and any pre-existing eye conditions. Subjects who underwent brain surgery, who have a neurological lesion, a psychiatric history or recurrent migraines that require medication will also be excluded from this study.

To minimize potential confounds, subjects with abnormal sleep/wake patterns will be excluded. They should report no sleep problems or shift work, or medications that could impair sleep, no illegal drugs or tobacco. Subjects will be in good health as assessed by medical history, interview and physical exam.

Subjects will be asked to:

Refrain from alcohol and caffeinated products for 1 day prior to the study;

Maintain their habitual bed times and wake-up times for 1 week prior to the study. A wrist-worn activity monitor (Actigraph[R], Precision Control Design, Inc., Fort Walton Beach, FL) may be used to confirm compliance with the latter instruction.

Exclusion criteria include:

Sleep disorder (reported or detected);

Psychopathology, personal or first-degree relative. (They are likely to place the subject at risk for an adverse consequence related to the extended wakefulness portion of the study);

Seizures or head injury with loss of consciousness greater than 5 minutes;

Substance dependence (diagnosable);

Smoking tobacco or psychotropic medications (currently);

Caffeine consumption of 300 mg or 2 ounces of alcohol on a regular daily consumption;

Cardiac, respiratory, or other medical condition that may affect cerebral metabolism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-06-28; Study Completion 2014-02-11

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Duyn, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bartels A, Zeki S. The chronoarchitecture of the human brain--natural viewing conditions reveal a time-based anatomy of the brain. Neuroimage. 2004 May;22(1):419-33. doi: 10.1016/j.neuroimage.2004.01.007. PMID 15110035
- [Background] Beckmann CF, Smith SM. Probabilistic independent component analysis for functional magnetic resonance imaging. IEEE Trans Med Imaging. 2004 Feb;23(2):137-52. doi: 10.1109/TMI.2003.822821. PMID 14964560
- [Background] Calhoun VD, Adali T, McGinty VB, Pekar JJ, Watson TD, Pearlson GD. fMRI activation in a visual-perception task: network of areas detected using the general linear model and independent components analysis. Neuroimage. 2001 Nov;14(5):1080-8. doi: 10.1006/nimg.2001.0921. PMID 11697939